CLINICAL TRIAL: NCT02204462
Title: FBnTP Positron Emission Mammography Imaging of Mitochondria Function - Breast Cancer
Brief Title: FBnTP Imaging of Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lock of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J13162; NA_00084913 (Other: JHM IRB)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: PET; Positron Emission Tomography; Breast Cancer; Imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — 18F-fluorobenzyl triphenyl phosphonium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Newly diagnosed breast cancer (Experimental): Patients with newly-diagnosed invasive and/or intraductal breast cancer detected by core needle or vacuum-assisted biopsy (i.e. index cancer). Patients will undergo FBnTP PET imaging for detection of malignant breast cancer.
  Interventions: Drug: FBnTP

INTERVENTIONS:
Drug: FBnTP — A PET imaging radiotracer
  Other Names: Fluorobenzyl triphenyl phosphonium

SUMMARY:
Our preclinical studies suggest the capacity of the positron emission tomography imaging agent 18F-fluorobenzyl triphenyl phosphonium (FBnTP) to detects early-stage small breast tumors (e.g., DCIS), and differentiates benign from malignant masses with better accuracy than that obtained by existing breast imaging tools.

DETAILED DESCRIPTION:
Breast cancer is the most widespread type of cancer among women in the USA, and the second leading cause of death. The National Cancer Institute estimates that in 2013, in the USA, 226,870 women will be diagnosed with breast cancer and 39,510 women will die of breast cancer, most of them of progressive metastatic disease. Early detection and treatment of the disease, when the tumor is still localized and at a high curability state, is the outmost important determinant of disease-free survival of breast cancer patients. Survival rate of women first diagnosed with pure early-stage noninvasive tumor (ductal carcinoma in situ- DCIS) is nearly 98%, which drops to 48% in patients with advanced disease.Yet, early detection of breast cancer is relatively poor. This is best exemplify by the astonishing percentage of benign biopsies; 80% of 1.7 million biopsies in the USA, at a cost of $3 billion; whereas, only small fraction (~20%) of newly diagnosed women are found to have pure DCIS.

Our preclinical studies suggest the capacity of the positron emission tomography (PET) imaging agent 18F-fluorobenzyl triphenyl phosphonium (FBnTP) to detects early-stage small breast tumors (e.g., DCIS), and differentiates benign from malignant masses with better accuracy than that obtained by existing breast imaging tools. Accordingly, the present protocol is designed to extend the preclinical findings into clinical studies in breast cancer women, and to assess the effectiveness of 18F-FBnTP in detecting breast malignant lesions, in comparison with magnetic resonance imaging and fluorodeoxyglucose PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with newly-diagnosed invasive and/or intraductal breast cancer detected by core needle or vacuum-assisted biopsy (i.e., index cancer)
* Age > 25 Ability and willingness to sign informed consent prior to any study procedure.
* Positive indication of disease on mammogram or MRI scan.
* Candidate for breast cancer surgery on the basis of recommendation of a breast cancer surgeon.
* Ability to undergo up to 90 minutes of PEM imaging.

Exclusion Criteria:

* Any active or chronic illness that, in the opinion of the investigators, would make the study unsafe or limit compliance with study procedures.
* Past or present history of active substance abuse (drug or alcohol).
* Inability to tolerate venous access.
* Pregnant females are excluded from this study. All females of child-bearing potential will undergo a serum pregnancy test within 48 hours prior to FBnTP administration.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Malignant breast cancer detection | Pre-treatment
  A feasibility study to assess the capacity of 18F-FBnTP PEM to detect and localize malignant breast lesions. Histopathology results will serve as reference standard.

SECONDARY OUTCOMES:
Imaging comparison | Pre-treatment
  To evaluate the concordance in detecting malignant breast lesions between FBnTP PEM and available diagnostic tests such as mammogram, 18F-FDG PEM or MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pomper, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
via manuscripts publication